CLINICAL TRIAL: NCT07307352
Title: 25010 - ABL90 FLEX PLUS - Precision Capillary Adult - Clinical Study Protocol
Status: Not yet recruiting | Type: Observational
Sponsor: Radiometer Medical ApS (Industry)
Responsible Party: Sponsor
Other Study IDs: 25010
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Diagnostic Tests
Keywords: ABL90

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: ABL90 FLEX PLUS analyser running SW3.5 MR2. — The ABL90 FLEX PLUS analyzer is a portable, automated analyzer that measures pH, blood gases, electrolytes, metabolites, and oximetry in whole blood - utilizing 3 measuring modes (syringe, short probe, and capillary mode) to measure samples from a syringe, test tube or a capillary tube. The analyzer provides results for 17 parameters in 35 seconds using 65 μL heparinized whole blood.

SUMMARY:
Conducting the ABL90 FLEX PLUS Clinical Precision Study for 15 Parameters in Adult Whole Blood is to validate performance claims for precision in heparinized whole blood for 15 parameters: pH, pCO2, pO2, cCa2+, cCl-, cK+, cNa+, cGlu, cLac, ctHb, sO2, FO2Hb, FMetHb, FCOHb, and FHHb, while being influenced by testing environment that is representative of intended use environment, site variability, and operator variability in a point-of-care (POC) setting.

The investigational device is the ABL90 FLEX PLUS (Figure 1) incl. consumables, running SW3.5 MR2, manufactured by Radiometer Medical ApS The study is being conducted in Denmark and in total, a minimum of 30 subjects are to be enrolled to provide successful measurement values from 2 sites.

DETAILED DESCRIPTION:
Adult Whole Blood is to validate performance claims for precision in heparinized whole blood for 15 parameters: pH, pCO2, pO2, cCa2+, cCl-, cK+, cNa+, cGlu, cLac, ctHb, sO2, FO2Hb, FMetHb, FCOHb, and FHHb, while being influenced by testing environment that is representative of intended use environment, site variability, and operator variability in a point-of-care (POC) setting.

Capillary blood collected into 2 capillary tubes from 2 distinct finger sticks will be measured on ABL90 FLEX PLUS in the Capillary mode (C65).

The study is designed to collect approximately 30 pairs of samples combined across sites.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be 18 years or older.
* Subjects must be able to understand given information and demonstrate willingness and ability to voluntarily give a signed, valid written informed consent to participate in the study.
* Subject evaluated as suitable according to the protocol to enroll in the study by the principal investigator or designee

Exclusion Criteria:

* Subject where sample collection is evaluated by principal investigator or designee to impose an unnecessary risk.
* Subject, with known pregnancy or breastfeeding.
* Subject, who has an invalid written informed consent or has withdrawn consent.
* Subjects who have been previously enrolled in the study.
* Subjects exposed to following substances within the last 72 hours:

  * Acetylsalicylic Acid Sodium Salt at dose equal or above 1 gram/day
  * N-acetylcysteine o Fluorescein dye o Patent Blue dye -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years old ) admitted to the hospital with low (moderate hypo), normal, or elevated (moderate hyper) concentrations of the 15 parameters covering the reportable range as much as possible.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-01-08 (Estimated); Primary Completion 2026-02-12 (Estimated); Study Completion 2026-02-12 (Estimated)

PRIMARY OUTCOMES:
Within sample precision for each parameter measured in capillary mode pooled across sites. | 1 hour
  Within sample precision of each parameter (pH, pCO2, pO2, cCa2+, cCl-, cK+, cNa+, cGlu, cLac, ctHb, sO2, FO2Hb, FMetHb, FCOHb and FHHb) using replicate measurements from heparinized whole blood samples measured by intended users in a POC setting.

SECONDARY OUTCOMES:
Within sample precision for each parameter measured in capillary mode per site, if applicable (at least 15 degrees of freedom shall be obtained for the estimate to be statistically meaningful). | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Klaus T Kristiansen, MD, Principal Investigator — Hvidovre Hospital, ICU; Lars Peter k Andersen, MD, Principal Investigator — Sjællands Universitetshospital Køge, Centre for Anaesthesiology
Locations (2):
- Denmark (2):
  - Hvidovre Hospital, Hvidovre
  - Sjællands Universitets Hospital Køge, Køge

IPD SHARING:
Plan to Share IPD: No
The clinical study results will be submitted to clinical trial.gov after study completion.